CLINICAL TRIAL: NCT02717403
Title: Phase 2 & Phase 3, Effects of Social Networking on Chronic Disease Management in Arthritis
Brief Title: Effects of Social Networking on Chronic Disease Management in Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Rheumatology Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-0349; 14038089 (Other Grant/Funding Number: Rheumatology Research Foundation); NCI-2016-00563 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-03-18; First posted 2016-03-23 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Chronic Disease Management; Rheumatoid Arthritis
Keywords: Chronic Disease Management; Rheumatoid Arthritis; Facebook; Social networking; Internet; Questionnaires; Surveys; Phone interview
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Surveys and Questionnaires; Media Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Facebook + Website Group (Experimental): Participants complete a self response electronic questionnaire at baseline. Participant shown how to access the Educational Website and the Facebook page on the internet about rheumatoid arthritis. Patients assessed at three and six months after baseline via email self response electronic questionnaires.
  Interventions: Behavioral: Questionnaires; Behavioral: Facebook; Behavioral: Educational Website
- Educational Website Group (Experimental): Participants complete a self response electronic questionnaire at baseline. Participant shown how to access the Educational Website on the internet about rheumatoid arthritis. Content includes the following: (i) a learning center; (ii) relevant links to other evidence-based web pages; (iii) news released by major rheumatology and dermatology organizations/societies; and (iv) chronic disease management strategies. Participants assessed at three and six months after baseline via email self response electronic questionnaires.
  Interventions: Behavioral: Questionnaires; Behavioral: Educational Website
- Pilot Testing Group (Experimental): Participants access the Educational Website and Facebook page about rheumatoid arthritis for a period of one week. After 1 week, research staff calls participant to obtain feedback about the websites. The interview will last approximately 30 minutes.
  Interventions: Behavioral: Facebook; Behavioral: Educational Website; Behavioral: Phone Interview

INTERVENTIONS:
Behavioral: Questionnaires — Participants complete a self response electronic questionnaire at baseline, and at three and six months.
  Other Names: Surveys
  Arms: Educational Website Group; Facebook + Website Group
Behavioral: Facebook — Participant accesses Facebook page regarding rheumatoid arthritis.
  Other Names: Social Media
  Arms: Facebook + Website Group; Pilot Testing Group
Behavioral: Educational Website — Participant accesses Educational Website on the internet about rheumatoid arthritis.
Behavioral: Phone Interview — Research staff calls participant to obtain feedback about the websites. The interview will last approximately 30 minutes.
  Arms: Pilot Testing Group

SUMMARY:
Objectives:

The overall goal of this study is to use the principles of chronic disease management to develop and test an online social networking intervention using the FB platform in a randomized controlled trial. Our specific objectives are as follows:

Aim 1: To develop and establish an independent closed community in FB for patients with rheumatoid arthritis, providing an educational platform for disease self-management and the potential for engaging in social networking with peers (Phase 2).

Objective 1. To beta test the features and navigation buttons and panels in the newly developed website and FB group.

Objective 2. To evaluate the contents, ease of use and satisfaction with the newly developed website and FB group by patient advocates (consultants to the study) who participate as members of the Facebook community.

Aim 2: To evaluate the efficacy of the FB community intervention combined with an educational website to improve patients' self-management (including knowledge, which is the primary outcome), decision making and patient-reported outcomes compared with the educational website alone (Phase 3). We hypothesize that participation in an online closed community offering evidence-based information combined with peer interaction and support will improve patients' knowledge.

DETAILED DESCRIPTION:
Pilot Testing Phase:

Five participants will be recruited to pilot test and give feedback on the control educational website and the FB community. Participants will have access to the educational website and FB, for a period of one week. The main purpose is to test ease of use and satisfaction with both platforms. After 1 week, research staff will call the participant to obtain feedback about the websites. The interview will last approximately 30 minutes and in the case the participant does not finish the interview, the investigators will conduct a follow-up phone interview.

Randomization Phase:

Participants will complete a self response electronic questionnaire at baseline. Participants then randomized into one of two arms: Intervention (FB + Website) and Control (Website alone). The participant will be shown how to access the website and the Facebook page on the internet about rheumatoid arthritis. Patients will be assessed at three and six months after baseline via email self response electronic questionnaires. This phase will recruit 220 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older (usability test and RCT)
2. Staff of the Department of General Internal Medicine (usability test)
3. Diagnosis of rheumatoid arthritis by a rheumatologist (RCT)
4. Ongoing or prior treatment with traditional disease-modifying anti-rheumatic drugs or biologic agents (RCT)
5. Adequate cognitive status as determined by a research coordinator at recruitment. To assess the participant's capacity to take part in the interview, the interviewer will note and comment on the participant's spontaneous speech and capacity to write date at the time of consent. Participants should be oriented to person, place, date, time, and events (RCT)
6. Living in the community (not institutionalized, etc. ) (RCT)
7. Able to communicate in English (RCT)
8. Use internet on average at-least once a week (RCT);
9. Disease duration 10 years or less (RCT)
10. Familiarity with and participation in social media (e.g. Facebook) (usability test and RCT)

Exclusion Criteria:

1. Participants not willing to complete interviews or survey instruments (usability test and RCT)
2. Hospitalized (RCT)
3. Patients who do not verbally, written, or electronically consent to participate (usability test and RCT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Participant Knowledge of Rheumatoid Arthritis assessed with the Patient Knowledge Questionnaire (PKQ-RA) | 6 months
  The Patient Knowledge Questionnaire (PKQ-RA) will measure this outcome.

SECONDARY OUTCOMES:
Control in Health Care Decisions assessed with the Control Preferences Scale (CPS-RA) | 6 months
  The Control Preferences Scale (CPS-RA) used to measure the degree of control an individual wants to assume while making decisions about their health care.

CONTACTS AND LOCATIONS:
Overall Officials: Angeles M. Lopez-Olivo, MD, PHD, MS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lopez-Olivo MA, Foreman JT, Leung C, Lin HY, Westrich-Robertson T, Hofstetter C, des Bordes JKA, Lyddiatt A, Leong A, Willcockson IU, Peterson SK, Suarez-Almazor ME. A randomized controlled trial evaluating the effects of social networking on chronic disease management in rheumatoid arthritis. Semin Arthritis Rheum. 2022 Oct;56:152072. doi: 10.1016/j.semarthrit.2022.152072. Epub 2022 Jul 16. PMID 35872394
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org